CLINICAL TRIAL: NCT07138833
Title: A Multicenter, Open-label, Single Group, Phase 4 Study to Evaluate Dimethyl Fumarate Enteric-coated Capsules in Relapsing Multiple Sclerosis (RMS)
Brief Title: A Phase IV Study of Dimethyl Fumarate Enteric-coated Capsules for Relapsing Multiple Sclerosis (RMS)
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Qilu Pharmaceutical (Hainan) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLG1031-401
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Relapsing Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dimethyl Fumarate Group (Experimental)
  Interventions: Drug: Dimethyl Fumarate Enteric-coated Capsules

INTERVENTIONS:
Drug: Dimethyl Fumarate Enteric-coated Capsules — Eligible 50 RMS patients will orally take dimethyl fumarate enteric-coated capsules during treatment, with an initial dose of 120 mg twice daily for 7 days, followed by a maintenance dose of 240 mg twice daily for 48 weeks

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety] in [subjects diagnosed with RMS according to the 2017 McDonald criteria, including clinically isolated syndrome (CIS), relapsing-remitting multiple sclerosis (RRMS), and active secondary progressive multiple sclerosis (SPMS).

The main questions it aims to answer are:

[Question 1] The efficacy of dimethyl fumarate enteric-coated capsules in the treatment of RMS.

[Question 2] The safety of dimethyl fumarate enteric-coated capsules in the treatment of RMS.

Participants will:

Eligible 50 RMS patients will orally take dimethyl fumarate enteric-coated capsules during treatment, with an initial dose of 120 mg twice daily for 7 days, followed by a maintenance dose of 240 mg twice daily for 48 weeks.

The annualized relapse rate (ARR) at Week 48 will be observed.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed RMS per the 2017 McDonald criteria, including clinically isolated syndrome (CIS), relapsing-remitting MS (RRMS), or active secondary progressive MS (SPMS)
* At least one documented relapse within 12 months prior to screening; plus evidence of MS-consistent lesions on prior brain MRI or gadolinium-enhancing (GdE) lesions on an MRI performed within 6 weeks before screening
* Expanded Disability Status Scale (EDSS) score between 0.0 and 5.0 (inclusive) at screening

Exclusion Criteria:

* History or current diagnosis of malignancy (except fully resected basal cell carcinoma), or uncontrolled severe diseases of major organ systems (e.g., cardiac, renal, hepatic, neurological [excluding multiple sclerosis]) that, in the investigator's assessment, pose a significant risk to the subject or could confound study results.
* Protocol-defined multiple sclerosis (MS) relapse within 30 days prior to screening, or failure to achieve clinical stability from a prior relapse.
* History of suicidal behavior within 5 years prior to screening. Suicidal ideation (indicated by a "Yes" response to Item 4 or 5 on the C-SSRS) within 6 months prior to screening.Subjects with a history of suicidal behavior occurring >5 years prior to screening require investigator assessment of eligibility.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Annualized Relapse Rate at Week 48 | 48 weeks
  The primary efficacy endpoint is the annualized relapse rate (ARR), calculated as total relapses divided by total patient-years of observation, measured at Week 48